CLINICAL TRIAL: NCT03268317
Title: Neuropsychiatric Adverse Effects in Patients With Chronic Hepatitis C Treated by Direct Acting Antiviral Drugs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariana Tharwat, Principle investigator, Assiut University
Other Study IDs: NAEIPWCHCTBDAAD
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic hepatitis C treated by DAAs: All subjects will be given the same treatment regimen which includes Sofosbuvir 400 mg orally/24 hours (pre-breakfast) and Daclatasvir 60 mg orally/24 hours after lunch with or without ribavirin for a total period of 12 weeks.

SUMMARY:
Neuropsychiatric adverse effects of direct acting antiviral drugs, especially Sofosbuvir and Daclatasvir combination therapy (with or without ribavirin) in patients with chronic hepatitis C , genotype four (the predominant genotype in Egypt).

DETAILED DESCRIPTION:
Treatment of hepatitis C virus, a virus infecting over one hundred seventy million worldwide, has evolved over the last two decades and moved from interferon-alpha monotherapy to pegylated interferon-alpha in combination with ribavirin therapy. Despite enhanced sustained virological response rates, psychiatric illness remains a barrier to widespread hepatitis C virus treatment uptake due to the neuropsychiatric risks associated with interferon-alpha.The next generation of hepatitis C virus therapeutic agents is direct acting antivirals that still require the use of interferon-ribavirin combination therapy.

Poorly managed psychiatric illness can lead not only to treatment discontinuation,but also poor adherence to treatment and serious psychiatric sequels, such as suicide.

Data on neuropsychiatric adverse effects of direct acting antivirals is limited and predominantly derived from landmark clinical trials for boceprevir and telaprevir.These first generation direct acting antivirals are currently not in use due to their multiple side effects ,the need for concomitant interferon-alpha ,and there wide drug-drug interactions. Recently the treatment of hepatitis C virus has undergone a paradigm shift with the introduction of the second generation of direct acting antivirals. This interferon-free modality has brought about exceptional cure rates with sustained virological response exceeding ninety hundred percent, with better tolerability, minimized side effects and short duration of treatment . Of the current hepatitis C virus treatment regimens, the combinations of Sofosbuvir plus daclatasvir have shown a high efficacy rate in achieving sustained virological response in genotype one patients.

To the investigators' knowledge, the development of neuropsychiatric side effects with the use of these second generation direct acting antivirals in absence of interferon therapy, as well as the impact of the expected high sustained virological response to therapy on the psychiatric condition of patients with chronic hepatitis C (in absence of cirrhosis) have not been studied. Therefore, the purpose of this work is to evaluate the neuropsychiatric adverse effects of direct acting antivirals,especially Sofosbuvir and Daclatasvir combination therapy (with or without ribavirin) in patients with chronic hepatitis C, genotype four (the predominant genotype in Egypt).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C only will be included.
* Patients who are eligible for treatment by DAAs only.

Exclusion Criteria:

* Cirrhotic patients will be excluded based on USS, APRI score index and FIB4 index.
* Hepatitis B infected patients will also be excluded.
* Patients with current or previous history of neuropsychiatric disorders will be excluded.
* Failure to obtain consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the Viral Hepatitis Clinic of Tropical Medicine Department, at Al-Rajhi Liver University Hospital Assiut, Egypt where these medications (DAAs) are available free for all insurance uncovered patients.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton anxiety scale (HAM-A) in patients with chronic hepatitis C treated by DAAs | 12 months
Hamilton depression scale (HAM-D) in patients with chronic hepatitis C treated by DAAs | 12 months

SECONDARY OUTCOMES:
EEG in patients with chronic hepatitis C treated by DAAs | 12 months
Visual evoked potential in patients with chronic hepatitis C treated by DAAs | 12 months

REFERENCES:
- [Background] Wasley A, Alter MJ. Epidemiology of hepatitis C: geographic differences and temporal trends. Semin Liver Dis. 2000;20(1):1-16. doi: 10.1055/s-2000-9506. PMID 10895428
- [Background] Dieperink E, Ho SB, Tetrick L, Thuras P, Dua K, Willenbring ML. Suicidal ideation during interferon-alpha2b and ribavirin treatment of patients with chronic hepatitis C. Gen Hosp Psychiatry. 2004 May-Jun;26(3):237-40. doi: 10.1016/j.genhosppsych.2004.01.003. PMID 15121353
- [Background] Ademmer K, Beutel M, Bretzel R, Jaeger C, Reimer C. Suicidal ideation with IFN-alpha and ribavirin in a patient with hepatitis C. Psychosomatics. 2001 Jul-Aug;42(4):365-7. doi: 10.1176/appi.psy.42.4.365. No abstract available. PMID 11496031
- [Background] Jacobson IM, McHutchison JG, Dusheiko G, Di Bisceglie AM, Reddy KR, Bzowej NH, Marcellin P, Muir AJ, Ferenci P, Flisiak R, George J, Rizzetto M, Shouval D, Sola R, Terg RA, Yoshida EM, Adda N, Bengtsson L, Sankoh AJ, Kieffer TL, George S, Kauffman RS, Zeuzem S; ADVANCE Study Team. Telaprevir for previously untreated chronic hepatitis C virus infection. N Engl J Med. 2011 Jun 23;364(25):2405-16. doi: 10.1056/NEJMoa1012912. PMID 21696307
- [Background] Poordad F, McCone J Jr, Bacon BR, Bruno S, Manns MP, Sulkowski MS, Jacobson IM, Reddy KR, Goodman ZD, Boparai N, DiNubile MJ, Sniukiene V, Brass CA, Albrecht JK, Bronowicki JP; SPRINT-2 Investigators. Boceprevir for untreated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1195-206. doi: 10.1056/NEJMoa1010494. PMID 21449783
- [Background] Sherman KE, Flamm SL, Afdhal NH, Nelson DR, Sulkowski MS, Everson GT, Fried MW, Adler M, Reesink HW, Martin M, Sankoh AJ, Adda N, Kauffman RS, George S, Wright CI, Poordad F; ILLUMINATE Study Team. Response-guided telaprevir combination treatment for hepatitis C virus infection. N Engl J Med. 2011 Sep 15;365(11):1014-24. doi: 10.1056/NEJMoa1014463. PMID 21916639
- [Background] Bacon BR, Gordon SC, Lawitz E, Marcellin P, Vierling JM, Zeuzem S, Poordad F, Goodman ZD, Sings HL, Boparai N, Burroughs M, Brass CA, Albrecht JK, Esteban R; HCV RESPOND-2 Investigators. Boceprevir for previously treated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1207-17. doi: 10.1056/NEJMoa1009482. PMID 21449784
- [Background] Gutierrez JA, Lawitz EJ, Poordad F. Interferon-free, direct-acting antiviral therapy for chronic hepatitis C. J Viral Hepat. 2015 Nov;22(11):861-70. doi: 10.1111/jvh.12422. Epub 2015 Jun 17. PMID 26083155
- [Background] Sulkowski MS, Gardiner DF, Rodriguez-Torres M, Reddy KR, Hassanein T, Jacobson I, Lawitz E, Lok AS, Hinestrosa F, Thuluvath PJ, Schwartz H, Nelson DR, Everson GT, Eley T, Wind-Rotolo M, Huang SP, Gao M, Hernandez D, McPhee F, Sherman D, Hindes R, Symonds W, Pasquinelli C, Grasela DM; AI444040 Study Group. Daclatasvir plus sofosbuvir for previously treated or untreated chronic HCV infection. N Engl J Med. 2014 Jan 16;370(3):211-21. doi: 10.1056/NEJMoa1306218. PMID 24428467